CLINICAL TRIAL: NCT03618732
Title: A Randomized Controlled Trial of Bilateral Movement-based Computer Games Training to Improve Motor Function of Upper Limb and Quality of Life in Sub-acute Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shatin Hospital (Other)
Responsible Party: Principal Investigator, Lam So Ling, Stefanie, Principal Investigator, Shatin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMRF02133096
Record Dates: First submitted 2017-10-06; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: stroke; upper limb; motor control; function; bilateral movement; virtual reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: stratified, single-blinded, intervention and controlled study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral movement-based computer training (Experimental): All subjects underwent 16 sessions of assigned treatment (2 times per week; for 8 weeks; 3 hours standardized rehabilitation program per visit) There was 1.5 hours standardized conventional physiotherapy training a 1.5 hours multi-disciplinary program which consisted of standardized occupational therapy, speech therapy and nursing care.
  Subjects in Intervention Group will be assigned an additional 30 minutes bilateral movement-based computer games(Able-X) training program of upper limb.
  Interventions: Other: Bilateral movement-based computer training
- Video-directed conventional training (Other): All subjects underwent 16 sessions of assigned treatment (2 times per week; for 8 weeks; 3 hours standardized rehabilitation program per visit) There was 1.5 hours standardized conventional physiotherapy training a 1.5 hours multi-disciplinary program which consisted of standardized occupational therapy, speech therapy and nursing care.
  Interventions: Other: Video-directed conventional training

INTERVENTIONS:
Other: Bilateral movement-based computer training
  Arms: Bilateral movement-based computer training
Other: Video-directed conventional training
  Arms: Video-directed conventional training

SUMMARY:
This study aims at investigating whether bilateral movement-based training with computer games could augment motor function of paretic upper limb and improve quality of life in sub-acute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45-85
* Diagnosis of ischaemic brain injury or intracerebral hemorrhage by MRI or computed tomography 1 week to 6 months after the onset of current stroke
* Scoring > 6 of 10 of Abbreviated Mental Test
* Ability of the paretic hand to hold the game controller (minimal control)
* Able to give informed consent of the study
* Can understand instructions given by English or Cantonese

Exclusion Criteria:

* Any additional medical, cardiovascular and orthopaedic condition that would hinder the proper assessment and treatment
* Having cardiac pacemaker
* Receptive dysphasia
* Undergoing drug studies or other clinical trials

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity Scores (FMA-UE scores) baseline to 4 weeks | Change from baseline to 4 weeks
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The FMA-UE scores measure motor impairment of upper extremity. The motor domain includes items assessing movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist and hand.
Fugl-Meyer Assessment-Upper Extremity Scores (FMA-UE scores) baseline to 8 weeks | Change from baseline to 8 weeks
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The FMA-UE scores measure motor impairment of upper extremity. The motor domain includes items assessing movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist and hand.
Fugl-Meyer Assessment-Upper Extremity Scores (FMA-UE scores) baseline to followup | Change from baseline to 12 weeks (4 weeks after training ended)
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The FMA-UE scores measure motor impairment of upper extremity. The motor domain includes items assessing movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist and hand.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) baseline to 4 weeks | Change from baseline to 4 weeks
  The Action Research Arm Test (ARAT) is an evaluative measure to assess specific changes in limb function among individuals who sustained cortical damage resulting in hemiplegia. It assesses a client's ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation.
Action Research Arm Test (ARAT) baseline to 8 weeks | Change from baseline to 8 weeks
  The Action Research Arm Test (ARAT) is an evaluative measure to assess specific changes in limb function among individuals who sustained cortical damage resulting in hemiplegia. It assesses a client's ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation.
Action Research Arm Test (ARAT) baseline to followup | Change from baseline to 12 weeks (4 weeks after training ended)
  The Action Research Arm Test (ARAT) is an evaluative measure to assess specific changes in limb function among individuals who sustained cortical damage resulting in hemiplegia. It assesses a client's ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation.
Short-Form Health Survey Hong Kong version (HK-SF-36) baseline to 4 weeks | Change from baseline to 4 weeks
  The Short-Form Health Survey (SF-36) is a widely used, generic, patient-report measure created to assess health-related quality of life (HRQOL) in the general population. SF-36 is the most commonly used generic instrument for measuring quality of life.
Short-Form Health Survey Hong Kong version (HK-SF-36) baseline to 8 weeks | Change from baseline to 8 weeks
  The Short-Form Health Survey (SF-36) is a widely used, generic, patient-report measure created to assess health-related quality of life (HRQOL) in the general population. SF-36 is the most commonly used generic instrument for measuring quality of life.
Short-Form Health Survey Hong Kong version (HK-SF-36) baseline to followup | Change from baseline to 12 weeks (4 weeks after training ended)
  The Short-Form Health Survey (SF-36) is a widely used, generic, patient-report measure created to assess health-related quality of life (HRQOL) in the general population. SF-36 is the most commonly used generic instrument for measuring quality of life.

IPD SHARING:
Plan to Share IPD: No